CLINICAL TRIAL: NCT03143595
Title: Cognitive Trajectories and Clinical Outcomes in Elderly Patients With Preoperative Cognitive Dysfunction
Brief Title: Clinical Outcomes in Elderly Patients With Preoperative Cognitive Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Jian-jun Yang, Professor, Zhongda Hospital
Other Study IDs: 20160530
Record Dates: First submitted 2017-04-26; First posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2016-05

CONDITIONS: Cognitive Decline; Age Problem; Outcome
Keywords: Preexisting cognitive impairment; Elderly; Outcomes
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Patients in this group have normal cognition as assessed by the validated Mini-Cog test before the elective operation.
- Impaired group: Patients in this group have impaired cognition as assessed by the validated Mini-Cog test before the elective operation.

SUMMARY:
Preexisting cognitive impairment, such as mild cognitive impairment, is common in many elderly patients who undergoing major surgeries. Accumulating evidence has demonstrated that preexisting cognitive impairment is associated with increased mortality, increased incidence of postoperative complications, decreased quality of life, and worse outcomes. However, few studies have evaluated the relationship between preexisting cognitive impairment and cognitive trajectories and clinical outcomes.

DETAILED DESCRIPTION:
Preexisting cognitive impairment is common in many elderly patients who undergoing major surgeries. The number of surgical procedures in the elderly will increase dramatically as a result of the increased elderly population in the future. It has been suggested that preexisting cognitive impairment is associated with increased incidence of postoperative complications, decreased quality of life, and increased mortality. Preoperative risk assessment is becoming increasingly important because preoperative risk stratification allows the clinical team to forecast postoperative outcomes. Currently, the most common strategy to identify high-risk patients before surgery is assessment of single end-organ function. This tactic is most widely recognized by the American Heart Association's guideline for cardiac evaluation, but is also well described for pulmonary, hepatic, and renal organ systems. Little is known about the effects of pre-existing cognitive (or brain) function (perhaps the most vital human organ) on postoperative outcomes. Therefore, the present study evaluated whether patients with pre-operative cognitive impairment would have a more precipitous drop in cognitive function and worse outcome in geriatric surgical patients.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion criteria were persons 65 years and older undergoing an elective operation on the general, noncardiac thoracic, urologic, and vascular surgical services.

Exclusion Criteria:

- Patients with vision or hearing impairment who could not visualize pictures or hear instructions associated with the delirium assessments and patients who could not provide informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients were 65 years and older undergoing an elective operation on the general, noncardiac thoracic, urologic, and vascular surgical services.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Cognition changes | 1 year
  Cognitive function was assessed at baseline before the elective operation and one year in all subjects using the Mini-Cog test by a member of a trained research team.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No